CLINICAL TRIAL: NCT00459251
Title: The Pharmacogenetics Study of Drug-Metabolising Enzyme Genetic Polymorphisms in Aboriginal and Minnan/Hakka Ethnic Groups in Taiwan
Brief Title: Pharmacogenetics Study in Taiwan's Ethnic Groups
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Department of Health (Ambiguous)
Other Study IDs: MMH-I-S-304
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Healthy
Keywords: N-acetyltransferase; Pharmacogenetics

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This main purpose of this study is to understand the difference and distribution of drug-metabolizing enzyme genetic polymorphisms among Taiwan ethnicities. The subjects of study include Atayal, Pawlan, Yami, Tsou, Ami, Minnan and Hakka. We anticipate establishing a reference for the clinical medication in various ethnic groups according to the difference and distribution of the genetic polymorphisms.

DETAILED DESCRIPTION:
It has been shown that the same medication causes different responses in different individuals. In addition to environments, diets, and physical conditions, the genetic variations play an important role in the various responses. For instant, genetic variations in drug-metabolism enzymes may be responsible to different abilities in drug metabolism. Some people have higher drug-metabolizing enzyme activity for certain drug and may need higher dose to reach the effective therapy; some are poor in metabolizing the same drug, and may cause adverse drug reactions. Genetic variation also may cause different functions of the cell transporters. The most notable example is that some tumor cells have a kind of transporters called p-glycoprotein which can pump out the anti-tumor drugs to extracellular, and it turns the tumor cells become resistant to the drugs. Hence, if we can elucidate the gene variation of each individual, we can give each individual different therapy based on their genetic variations. This approach is called 「individualized medicine」.

In order to reach the goal of individualized medicine, many studies have been focused on drug-metabolizing enzyme genetic variations between races or ethnicities. Especially, single nucleotide polymorphism provides a very important basis to clinical medication. N- acetyltransferase 2 (NAT2) is one kind of drug-metabolizing enzymes and its single nucleotide polymorphisms have remarkable effect on drug-metabolism. Only 10~30 % are slow acetylators in Asian population, but 40~70% are found in Caucasian population. Cytochrome P450 (CYP450,CYP) is another important drug-metabolizing enzyme family. Among the family, the CYP2C9, CYP2C19, and CYP2D6 play key roles on drug metabolism. Many literatures showed that all the three enzymes have various distributions of SNPs in different races. It indicates that different races may have different abilities in drug-metabolizing enzymes. Therefore, it is important to provide a strategy to overcome the difficulties in individualized medicine.

In the previous studies, scientists often take Chinese as the representatives of Asian people and the Minnan/ Hakka or so-called Han people as the subjects when study the Taiwan ethnicity. The genetic variations in the Taiwan aborigines are poorly investigated. It has been showed that remarkable genetic variations in human leukocyte antigen (HLA) between Taiwan aborigines and Minnan/ Hakka by Lin ML and her colleagues. They are highly homogenous within each tribe, but diversified among the different tribes due to long-term isolation. Therefore, we expect to establish a database of genetic variations in drug-metabolism enzymes among these groups in order to use as the basis for clinical medication. This study includes seven groups, and each of them has 50 independent samples for drug-metabolizing enzyme genetic polymorphism analysis. The important enzymes, CYP2C9, CYP2C19, CYP2D6 and NAT2, etc., are studied in this project. ABI 7900HT instrument and traditional polymerase chain reaction (PCR) - restriction fragment length polymorphism (RFLP) both are used for SNPs analysis, and gene sequence also would be used to confirm the results.

ELIGIBILITY:
Inclusion Criteria:

* This study includes seven groups, and each of them has 50 independent samples for drug-metabolizing enzyme genetic polymorphism analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2006-12; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiuan Shen, Ph.D., Principal Investigator — School of Pharmacy, National Taiwan University
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Chu CC, Lin M, Nakajima F, Lee HL, Chang SL, Juji T, Tokunaga K. Diversity of HLA among Taiwan's indigenous tribes and the Ivatans in the Philippines. Tissue Antigens. 2001 Jul;58(1):9-18. doi: 10.1034/j.1399-0039.2001.580102.x. PMID 11580850